CLINICAL TRIAL: NCT02942212
Title: Health Literacy and Smoking Cessation in Low-SES Diverse Smokers - Project HALT II
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No activties have occurred and no participants have enrolled in this protocol
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-0267; NCI-2018-02698 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-10-20; First posted 2016-10-24 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; Nicotine patch; Nicoderm Committed Quitters; CQ; Nicoderm CQ; Questionnaires; Surveys; Interviews; Breath tests
MeSH Terms: conditions — Smoking Cessation | interventions — Surveys and Questionnaires; Tobacco Use Cessation Devices; Nicotine; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Project HALT II: In-Depth Interviews (Experimental): Participants complete a computerized questionnaire to assess demographics and smoking history.
  Participants take part in individual in-depth interviews discussing smoking history, attempts to quit, and suggestions for smoking cessation program.
  Interventions: Behavioral: Questionnaire; Behavioral: In-Depth Interviews
- Project HALT II: Standard Treatment (ST) (Active Comparator): Participants complete a computerized questionnaire to assess demographics and smoking history at baseline.
  Participants complete a breath test to assess the amount of cigarette smoke inhaled at baseline, weekly during study, and at 3 month follow up.
  Participants receive a 6-week supply of nicotine patches and instructions on how to use them. Participants receive brief advice to quit smoking. Participants receive phone counseling for support in quitting smoking (5 sessions over the course of 6 weeks) with a counselor at the Texas Quitline.
  Participants complete self assessment questionnaires the week before quitting smoking, the day that they quit, and 1, 2, and 4 weeks after quitting, and at 3 month follow up.
  Interventions: Behavioral: Questionnaire; Other: Breath Test; Drug: Nicotine Patches; Behavioral: Advice plus Phone Counseling; Behavioral: Self Assessment Questionnaires
- Project HALT II: Tailored Treatment (HALT) (Experimental): Participants complete a computerized questionnaire to assess demographics and smoking history at baseline.
  Participants complete a breath test to assess the amount of cigarette smoke inhaled at baseline, weekly during study, and at 3 month follow up.
  Participants receive a 6-week supply of nicotine patches and instructions on how to use them. Participants receive brief advice to quit smoking. Participants scheduled to attend 5 individual, in-person smoking cessation treatment counseling sessions.
  Participants complete self assessment questionnaires the week before quitting smoking, the day that they quit, and 1, 2, and 4 weeks after quitting, and at 3 month follow up.
  Interventions: Behavioral: Questionnaire; Other: Breath Test; Drug: Nicotine Patches; Behavioral: Advice plus Counseling Sessions; Behavioral: Self Assessment Questionnaires

INTERVENTIONS:
Behavioral: Questionnaire — Participants complete a computerized questionnaire to assess demographics and smoking history.
  Other Names: Survey
Behavioral: In-Depth Interviews — Participants take part in individual in-depth interviews discussing smoking history, attempts to quit, and suggestions for smoking cessation program. The interview should last 30-45 minutes and is audio-recorded.
  Arms: Project HALT II: In-Depth Interviews
Other: Breath Test — Participants complete a breath test to assess the amount of cigarette smoke inhaled at baseline, weekly during study, and at 3 month follow up.
  Arms: Project HALT II: Standard Treatment (ST); Project HALT II: Tailored Treatment (HALT)
Drug: Nicotine Patches — Participants receive a 6-week supply of nicotine patches and instructions on how to use them. Patch therapy for participants who smoke >10 cigarettes/day consists of 4 weeks of 21 mg patches, 1 week of 14 mg patches, and 1 week of 7 mg patches. Patch therapy for participants who smoke 5-10 cigarettes/day consists of 4 weeks of 14 mg patches and 2 weeks of 7 mg patches.
  Other Names: Nicoderm Committed Quitters (CQ); Nicoderm CQ
  Arms: Project HALT II: Standard Treatment (ST); Project HALT II: Tailored Treatment (HALT)
Behavioral: Advice plus Phone Counseling — Participants receive brief advice to quit smoking, as well as phone counseling for support in quitting smoking (5 sessions over the course of 6 weeks) with a counselor at the Texas Quitline.
  Arms: Project HALT II: Standard Treatment (ST)
Behavioral: Advice plus Counseling Sessions — Participants receive brief advice to quit smoking, as well as 5 individual, in-person smoking cessation treatment counseling sessions.
  Arms: Project HALT II: Tailored Treatment (HALT)
Behavioral: Self Assessment Questionnaires — Participants complete self assessment questionnaires the week before quitting smoking, the day that they quit, and 1, 2, and 4 weeks after quitting, and at 3 month follow up.
  Other Names: Surveys
  Arms: Project HALT II: Standard Treatment (ST); Project HALT II: Tailored Treatment (HALT)

SUMMARY:
In-Depth Interviews:

The goal of this research study is to learn about ways to help people might have trouble understanding health information quit smoking.

Pilot Study:

The goal of this research study is to test 2 different approaches, Standard Treatment (ST) and Helping Adults with Health Literacy Trouble (HALT) tailored treatment, for helping smokers who might have trouble understanding health information with quitting smoking.

DETAILED DESCRIPTION:
In-Depth Interviews:

Study Visit:

If participant is eligible and agrees to take part, the following will occur at their visit:

Questionnaire:

Participant will complete a questionnaire on a computer that will include questions about their thoughts about smoking, their smoking history, their ability to understand health information, and basic questions about their age, education, and income. This may take up to 45 minutes to complete.

Individual In-Depth Interviews:

After completing the questionnaire, participant will take part in an individual, in-depth interview. As part of the interview, the study chair will ask participant about their smoking, any previous attempts at quitting, and what they would like to see included as part of a program to help smokers like them with quitting smoking.

The interview should last 30-45 minutes and will be audio-recorded. No identifying information will be included in recorded interviews (participant's name will not be used). Recordings will be transcribed (written down). Audio recordings will be permanently deleted within a year after the completion of data collection.

Length of Study Participation:

It may take up to 2 hours to complete this visit. Participation in this study will be over after participant completes the interview.

Pilot Study:

Baseline Visit:

If participant is eligible and agrees to take part in this study, the following will occur when they start the study (also called a baseline visit):

* Participant will complete a questionnaire on the computer that will include questions about their feelings, mood, health, thoughts about smoking, thoughts about quitting smoking, and their smoking history. It will also include questions about participant's age, education, and income. This may take up to 1 hour to complete.
* Participant will complete a breath test to help the research team learn about the amount of cigarette smoke they inhale. The breath test uses a disposable cardboard tube attached to a machine, and participant will be asked to blow a long, slow, steady breath into it.
* Participant will then be randomly assigned (as in the flip of a coin) into 1 of 2 study groups (explained below). This is done because no one knows if one study group is better, the same, or worse than the other group. There is an equal chance of being assigned to either group.

Study Groups:

If participant is in Group 1 (ST):

* Participant will receive a 6-week supply of nicotine patches and instructions on how to use them.
* Participant will receive brief advice to quit smoking.
* Participant will receive phone counseling for support in quitting smoking (5 sessions over the course of 6 weeks) with a counselor at the Texas Quitline, an organization that helps people quit smoking. Counseling is designed to help participant to improve their problem-solving and coping skills, and plan for quitting smoking. Calls are expected to last up to 45 minutes.

If participant is in Group 2 (HALT):

* Participant will receive a 6-week supply of nicotine patches and instructions on how to use them.
* Participant will receive brief advice to quit smoking.
* Participant will receive 5 individual, in-person counseling sessions for support in quitting smoking. Sessions are designed to help participant to improve their problem-solving and coping skills, overcome barriers to quitting smoking, and plan for quitting smoking. These sessions will take place at either of Literacy Advance's 2 main campuses over 6 weeks. Participant will attend sessions the week before they quit smoking, on the day that they quit, and 1, 2, and 4 weeks after quitting. Each of these sessions will last about 45 minutes.

Weekly In-Person Visits (Groups 1 and 2):

Participant will complete questionnaires in person and at Literacy Advance over 6 weeks (the week before they quit smoking, on the day that they quit, and 1, 2, and 4 weeks after quitting). These questionnaires will ask about participant's current smoking, motivation to quit smoking, confidence for quitting, stress, and emotions/mood. Participant will also complete a breath test to help researchers learn about the amount of cigarette smoke participant inhales. This should take about 30 minutes to complete.

3-Month In-Person Follow-Up Visit (Groups 1 and 2): Eight (8) weeks after the last counseling session (or 3 months after beginning the study), participant will attend an in-person, follow-up visit in which they will complete questionnaires and a breath test to help the researchers learn about the amount of cigarette smoke participant inhales. This should take about 30 minutes to complete.

Length of Study:

If participant does not quit smoking on their "Quit Day" (Week 0), they may continue participating in the study and may select another "Quit Day."

Participant will take part in the study for up to 3 months. Participation will be over when participant completes the study visit at Month 3.

This is an investigational study. The nicotine patch is FDA approved and commercially available.

Up to 50 participants will take part in this pilot study. Up to 80 participants overall will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. (IN-DEPTH INTERVIEWS - INCLUSION CRITERIA; 2-6)
2. Age 25-65 years
3. Current smoker (>/= 5 cigarettes/day for the last year)
4. Limited or marginal HL (total score </=6 on the CHEW Questionnaire)
5. Have a home address where information can be mailed and a working telephone
6. English speaker
7. Currently attending Adult Basic Education (ABE) classes at Literacy Advance of Houston
8. (PILOT STUDY - INCLUSION CRITERIA; 8-13)
9. Age 25-65 years
10. Current smoker (>/= 5 cigarettes/day for the last year; biochemically verified with expired carbon monoxide (CO) reading of >/=8 parts per million [ppm])
11. Limited or marginal HL (total score </=6 on the CHEW Questionnaire)
12. Motivated to quit smoking within the next 30 days
13. Have a home address where information can be mailed and a working telephone
14. English speaker
15. Currently attending Adult Basic Education (ABE) classes at Literacy Advance of Houston

Exclusion Criteria:

1. (IN-DEPTH INTERVIEWS - EXCLUSION CRITERIA; 2-5)
2. Regular use of tobacco products other than cigarettes
3. Current use of tobacco cessation medications
4. Pregnancy or lactation
5. Enrolled in another smoking cessation study/program
6. (PILOT STUDY - EXCLUSION CRITERIA; 7-12)
7. Contraindication for nicotine patch
8. Regular use of tobacco products other than cigarettes
9. Current use of tobacco cessation medications
10. Pregnancy or lactation
11. A household member is enrolled in the study
12. Enrolled in another smoking cessation study/program

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Efficacy of Helping Adults with Health Literacy Trouble (HALT) versus Standard Treatment (ST) in Facilitating Abstinence from Smoking in Low Health Literacy (HL) Smokers | 3 months
  Efficacy defined as the proportion of participants who successfully quit smoking.

CONTACTS AND LOCATIONS:
Overall Officials: Diana S. Hoover, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- Literacy Advance of Houston, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org